CLINICAL TRIAL: NCT03834519
Title: A Phase 3, Randomized Open-label Study of Pembrolizumab (MK-3475) Plus Olaparib Versus Abiraterone Acetate or Enzalutamide in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) Who Are Unselected for Homologous Recombination Repair Defects and Have Failed Prior Treatment With One Next-generation Hormonal Agent (NHA) and Chemotherapy (KEYLYNK-010)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Olaparib Versus Abiraterone Acetate or Enzalutamide in Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-7339-010/KEYLYNK-010)
Acronym: KEYLYNK-010
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7339-010; MK-7339-010 (Other: MSD); KEYLYNK-010 (Other: MSD); 2018-004118-16 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Prostatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; olaparib; Abiraterone Acetate; Prednisone; enzalutamide; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Olaparib (Experimental): Participants will receive olaparib 600 mg as two 150 mg oral tablets twice daily (BID) continuously until progression PLUS on Day 1 of each 21-day cycle, pembrolizumab 200 mg by intravenous (IV) infusion for up to 35 cycles (approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Olaparib
- Next-generation Hormonal Agent Monotherapy (NHA) (Active Comparator): Participants will receive a single NHA, which will be either abiraterone acetate (participants previously treated with enzalutamide) 1000 mg as two 500 mg or four 250 mg oral tablets once daily (QD) PLUS prednisone or prednisolone 10 mg as one 5 mg tablet BID until progression OR enzalutamide (participants previously treated with abiraterone acetate) 160 mg as four 40 mg oral tablets or capsules OR two 80 mg tablets QD until progression.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Enzalutamide; Drug: Prednisolone

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Olaparib
Drug: Olaparib — Oral tablets
  Other Names: MK-7339; AZD-2281; LYNPARZA®
  Arms: Pembrolizumab + Olaparib
Drug: Abiraterone acetate — Oral tablets
  Other Names: ZYTIGA®; CB-7630; JNJ-212082
  Arms: Next-generation Hormonal Agent Monotherapy (NHA)
Drug: Prednisone — Oral tablets
  Arms: Next-generation Hormonal Agent Monotherapy (NHA)
Drug: Enzalutamide — Oral tablets or oral capsules
  Other Names: XTANDI®; MDV-3100; ASP-9785
  Arms: Next-generation Hormonal Agent Monotherapy (NHA)
Drug: Prednisolone — Oral tablets
  Arms: Next-generation Hormonal Agent Monotherapy (NHA)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of the polyadenosine 5'-diphosphoribose poly (ADP-ribose) polymerase (PARP) inhibitor olaparib and pembrolizumab in the treatment of participants with mCRPC who have failed to respond to either abiraterone acetate or enzalutamide (but not both) and to chemotherapy.

The primary study hypotheses are that the combination of pembrolizumab plus olaparib is superior to abiraterone acetate or enzalutamide with respect to:

1. Overall Survival (OS) and
2. Radiographic progression-free survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 as assessed by blinded independent central review (BICR)

As of Amendment 06, the Data Monitoring Committee (DMC) is no longer applicable. Participants still on treatment may have the option to continue receiving study intervention or SOC if they are deriving clinical benefit, until criteria for discontinuation are met. Participants who are still on study treatment and deriving clinical benefit will no longer have tumor response assessments by BICR. However, local tumor imaging assessments should continue per standard of care (SOC) schedule. In addition, electronic patient-reported outcome (ePRO) assessments will no longer be performed and biomarker samples will no longer be collected.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while receiving androgen deprivation therapy (or post bilateral orchiectomy) within 6 months before screening
* Has current evidence of metastatic disease documented by bone lesions on bone scan and/or soft tissue disease shown by computed tomography/magnetic resonance imaging (CT/MRI)
* Has received prior treatment with abiraterone acetate OR enzalutamide, but not both

  * Have disease that progressed during or after treatment with abiraterone acetate for either metastatic hormone-sensitive prostate cancer (mHSPC) or mCRP or enzalutamide for mCRPC for at least 8 weeks (at least 14 weeks for participants with bone progression)
  * Participants that received abiraterone acetate for mHSPC may not have received abiraterone acetate or enzalutamide for mCRPC
* Have received docetaxel chemotherapy regimen for metastatic castration-resistant prostate cancer (mCRPC) and have had progressive disease during or after treatment with docetaxel
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM)
* If receiving bone resorptive therapy, including but not limited to bisphosphonates or denosumab, must have been receiving stable doses before randomization
* Must agree to refrain from donating sperm during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention PLUS be abstinent from heterosexual intercourse OR must agree to use contraception unless confirmed to be azoospermic
* Contraception use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirement above, the local label requirements are to be followed.
* Has provided tumor tissue from a fresh core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated. Samples from tumors progressing at a prior site of radiation are allowed. Participants with bone-only or bone-predominant disease may provide a bone biopsy sample
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis requiring steroids, or has current pneumonitis
* Has known active human immunodeficiency virus (HIV), hepatitis B virus (e.g., hepatitis B surface antigen reactive) or hepatitis C virus (HCV) infection (e.g., HCV RNA [qualitative] is detected)
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of seizure or any condition that may predispose to seizure
* Has a history of loss of consciousness within 12 months of screening
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has (≥Grade 3) hypersensitivity to pembrolizumab and/or any of its excipients
* Has known hypersensitivity to the components or excipients in olaparib, abiraterone acetate, prednisone or prednisolone, or enzalutamide
* Has symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease)
* Has received an anticancer monoclonal antibody (mAb) before randomization
* Has received prior treatment with olaparib or any other PARP inhibitor
* Has received prior treatment with apalutamide or darolutamide
* Has received prior treatment with enzalutamide or apalutamide for metastatic hormone-sensitive prostate cancer
* Has used herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA (e.g., saw palmetto) before the date of randomization
* Has received prior treatment with radium or other therapeutic radiopharmaceuticals for prostate cancer
* Has received prior treatment with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, or CD137)
* Is currently receiving either strong or moderate inhibitors of cytochrome P450 [CYP] (CYP3A4) that cannot be discontinued for the duration of the study
* Has received a previous allogenic bone marrow transplant or double umbilical cord transplantation (dUCBT) or a solid organ transplant
* Has received a live vaccine within 30 days prior to the date of randomization
* Is currently participating in or has participated in a study of an investigational agent, or has used an investigational device, within 4 weeks before the date of randomization
* Has a bone "superscan"
* Is expecting to father children within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2024-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (193):
- United States (29):
  - St. Joseph Heritage Healthcare ( Site 0069), Fullerton, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0081), Los Angeles, California
  - Sibley Memorial Hospital ( Site 0096), Washington D.C., District of Columbia
  - Georgia Cancer Center at Augusta University ( Site 0026), Augusta, Georgia
  - Quincy Medical Group ( Site 0021), Quincy, Illinois
  - Tulane Cancer Center ( Site 0066), New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 0005), Baltimore, Maryland
  - Chesapeake Urology Research Associates ( Site 0076), Towson, Maryland
  - Beth Israel Deaconess Medical Ctr. ( Site 0093), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0033), Boston, Massachusetts
  - UMass Memorial Medical Center ( Site 0053), Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute ( Site 0077), Detroit, Michigan
  - Henry Ford Health System ( Site 0039), Detroit, Michigan
  - St. Vincent Frontier Cancer Center ( Site 0016), Billings, Montana
  - Nebraska Cancer Specialists ( Site 0034), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada ( Site 0092), Las Vegas, Nevada
  - University of New Mexico Cancer Center ( Site 0048), Albuquerque, New Mexico
  - Memorial Medical Center ( Site 0095), Las Cruces, New Mexico
  - Associated Medical Professionals of NY ( Site 0060), Syracuse, New York
  - Duke Cancer Center Cary ( Site 0010), Cary, North Carolina
  - Gabrail Cancer Center-Research ( Site 0097), Canton, Ohio
  - The Urology Group- Cincinnati ( Site 0094), Cincinnati, Ohio
  - University Hospitals of Cleveland Seidman Cancer Center ( Site 0036), Cleveland, Ohio
  - Carolina Urologic Research Center ( Site 0070), Myrtle Beach, South Carolina
  - Huntsman Cancer Institute ( Site 0002), Salt Lake City, Utah
  - Virginia Cancer Institute ( Site 0052), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0086), Roanoke, Virginia
  - Seattle Cancer Care Alliance ( Site 0079), Seattle, Washington
  - Froedtert and Medical College of Wisconsin ( Site 0045), Milwaukee, Wisconsin
- Argentina (8):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 1013), Berazategui, Buenos Aires
  - Centro de Diagnostico Urologico ( Site 1008), Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 1006), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 1002), Rosario, Santa Fe Province
  - Instituto de Investigaciones Metabolicas ( Site 1011), Buenos Aires
  - Hospital Aleman ( Site 1004), Buenos Aires
  - Instituto Medico Alexander Fleming ( Site 1010), Buenos Aires
  - CEMAIC ( Site 1014), Córdoba
- Australia (10):
  - St. Vincent's Hospital ( Site 0158), Darlinghurst, New South Wales
  - Macquarie University ( Site 0151), Macquarie University, New South Wales
  - Port Macquarie Base Hospital ( Site 0153), Port Macquarie, New South Wales
  - Calvary Mater Newcastle ( Site 0148), Waratah, New South Wales
  - Southern Medical Day Care Centre ( Site 0160), Wollongong, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0155), Herston, Queensland
  - John Flynn Hospital & Medical Centre ( Site 0164), Tugun, Queensland
  - Box Hill Hospital ( Site 0146), Box Hill, Victoria
  - Peter MacCallum Cancer Centre ( Site 0152), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0162), Murdoch, Western Australia
- Austria (4):
  - Medizinische Universitat Graz ( Site 0374), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 0373), Linz, Upper Austria
  - SCRI-CCCIT GesmbH ( Site 0371), Salzburg
  - Medizinische Universitaet Wien ( Site 0375), Vienna
- Brazil (6):
  - Hospital de Caridade de Ijui ( Site 1038), Ijuí, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 1021), Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 1035), Itajaí, Santa Catarina
  - Hospital de Base de Sao Jose de Rio Preto ( Site 1022), São José do Rio Preto, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer ( Site 1040), São Paulo, São Paulo
  - A.C. Camargo Cancer Center ( Site 1026), São Paulo
- Canada (10):
  - Cross Cancer Institute ( Site 0110), Edmonton, Alberta
  - BC Cancer-Kelowna - Sindi Ahluwalia Hawkins Centre ( Site 0113), Kelowna, British Columbia
  - BC Cancer-Vancouver Center ( Site 0112), Vancouver, British Columbia
  - Nova Scotia Health Authority QEII-HSC ( Site 0114), Halifax, Nova Scotia
  - William Osler Health System (Brampton Civic Hospital) ( Site 0121), Brampton, Ontario
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0116), Hamilton, Ontario
  - Princess Margaret Cancer Centre ( Site 0107), Toronto, Ontario
  - CHUQ-Univ Laval-Hotel Dieu de Quebec ( Site 0103), Québec, Quebec
  - CIUSSS du Bas Saint Laurent - Hopital Regional de Rimouski ( Site 0102), Rimouski, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0105), Sherbrooke, Quebec
- Chile (5):
  - Fundacion Arturo Lopez Perez ( Site 1049), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1047), Santiago, Region M. de Santiago
  - Bradford Hill Centro de Investigaciones Clinicas ( Site 1044), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1041), Temuco, Región de la Araucanía
  - Rey y Oreilly Limitada ( Site 1048), Temuco, Región de la Araucanía
- France (19):
  - C.H. de Saint Quentin ( Site 0481), Saint-Quentin, Aisne
  - Clinique Sainte Anne ( Site 0431), Strasbourg, Alsace
  - Centre Jean Perrin ( Site 0434), Clermont-Ferrand, Auvergne
  - Institut Paoli Calmettes ( Site 0419), Marseille, Bouches-du-Rhone
  - CHU de Brest -Site Hopital Morvan ( Site 0441), Brest, Brittany Region
  - CHU Jean Minjoz ( Site 0423), Besançon, Doubs
  - Institut Bergonie ( Site 0421), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0418), Toulouse, Haute-Garonne
  - Hopital Foch ( Site 0428), Suresnes, Hauts-de-Seine
  - Institut Regional du Cancer de Montpellier - ICM ( Site 0443), Montpellier, Herault
  - Institut De Cancerologie De L Ouest ( Site 0448), Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Regional du Orleans ( Site 0430), Orléans, Loiret
  - Centre D Oncologie de Gentilly ( Site 0432), Nancy, Meurthe-et-Moselle
  - Centre Leon Berard ( Site 0422), Lyon, Rhone
  - C.H.U. Lyon Sud ( Site 0436), Pierre-Bénite, Rhone
  - CHU Amiens Picardie Site Sud Amiens ( Site 0438), Amiens, Somme
  - Institut Gustave Roussy ( Site 0416), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 0447), Avignon, Vaucluse
  - Institut Mutualiste Montsouris ( Site 0446), Paris
- Germany (11):
  - Universitaetsklinikum Freiburg - Medizinische Klinik ( Site 0304), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum in Mannheim ( Site 0314), Mannheim, Baden-Wurttemberg
  - Studienpraxis Urologie ( Site 0309), Nürtingen, Baden-Wurttemberg
  - Universitaetsklinik fuer Urologie ( Site 0307), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 0303), Erlangen, Bavaria
  - Klinikum Rechts der Isar ( Site 0300), Munich, Bavaria
  - Universitaetsklinik der Paracelsus Medizinischen Privatuniversitaet ( Site 0318), Nuremberg, Bavaria
  - Universitaetsklinikum Duesseldorf ( Site 0306), Düsseldorf, North Rhine-Westphalia
  - Krankenhaus der Barmherzigen Brueder Trier ( Site 0310), Trier, Rhineland-Palatinate
  - Universitaetsklinikum Jena ( Site 0305), Jena, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0301), Berlin
- Ireland (2):
  - Tallaght University Hospital ( Site 0730), Dublin
  - Mid Western Cancer Centre ( Site 0728), Limerick
- Israel (9):
  - Ha Emek Medical Center ( Site 0548), Afula
  - Soroka Medical Center ( Site 0549), Beersheba
  - Assaf Harofe ( Site 0547), Be’er Ya‘aqov
  - Rambam Medical Center ( Site 0543), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0546), Jerusalem
  - Meir Medical Center ( Site 0544), Kfar Saba
  - Rabin Medical Center ( Site 0545), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0541), Ramat Gan
  - Sourasky Medical Center ( Site 0542), Tel Aviv
- Italy (9):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 0462), Meldola, Emilia-Romagna
  - Istituto Clinico Humanitas Research Hospital ( Site 0452), Rozzano, Lombardy
  - Medical Oncology Ospedale San Donato ( Site 0461), Arezzo
  - Policlinico S.Orsola-Malpighi ( Site 0453), Bologna
  - Azienda Ospedaliera Cannizzaro ( Site 0458), Catania
  - Azienda Ospedaliera San Camillo Forlanini ( Site 0455), Roma
  - Fondazione Policlinico Universitario A. Gemelli ( Site 0463), Roma
  - Azienda Ospedaliera Santa Maria Terni ( Site 0456), Terni
  - Presidio Ospedaliero Santa Chiara ( Site 0451), Trento
- Japan (25):
  - Fujita Health University Hospital ( Site 0724), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 0702), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 0703), Sakura, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0716), Matsuyama, Ehime
  - Kobe City Medical Center General Hospital ( Site 0726), Kobe, Hyōgo
  - Kanazawa University Hospital ( Site 0701), Kanazawa, Ishikawa-ken
  - Kitasato University Hospital ( Site 0705), Sagamihara, Kanagawa
  - Yokohama City University Medical Center ( Site 0706), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 0715), Kashihara, Nara
  - Kindai University Hospital ( Site 0714), Sayama, Osaka
  - Osaka University Hospital ( Site 0713), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 0708), Hidaka, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 0707), Koshigaya, Saitama
  - Fuji City General Hospital ( Site 0725), Fuji, Shizuoka
  - Hamamatsu University Hospital ( Site 0720), Hamamatsu, Shizuoka
  - Yamaguchi University Hospital ( Site 0717), Ube, Yamaguchi
  - Chiba Cancer Center ( Site 0704), Chiba
  - Kyushu University Hospital ( Site 0718), Fukuoka
  - University of Miyazaki Hospital ( Site 0721), Miyazaki
  - Nagano Municipal Hospital ( Site 0723), Nagano
  - Nagasaki University Hospital ( Site 0719), Nagasaki
  - Osaka International Cancer Institute ( Site 0722), Osaka
  - Toranomon Hospital ( Site 0711), Tokyo
  - Nippon Medical School Hospital ( Site 0709), Tokyo
  - Keio University Hospital ( Site 0710), Tokyo
- Netherlands (9):
  - Radboud University Medical Center ( Site 0470), Nijmegen, Gelderland
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 0480), Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum ( Site 0479), Amsterdam, North Holland
  - Spaarne Ziekenhuis ( Site 0473), Hoofddorp, North Holland
  - Ziekenhuisgroep Twente ( Site 0469), Hengelo, Overijssel
  - Medisch Centrum Leeuwarden ( Site 0477), Leeuwarden, Provincie Friesland
  - Haaglanden MC - locatie Antoniushove ( Site 0471), Leidschendam, South Holland
  - Erasmus MC ( Site 0475), Rotterdam, South Holland
  - Franciscus Gasthuis en Vlietland ( Site 0489), Schiedam, South Holland
- Auckland City Hospital ( Site 0193), Auckland, New Zealand
- Russia (10):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 0565), Chelyabinsk, Chelyabinsk Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0585), Krasnoyarsk, Krasnoyarsk Krai
  - Russian Scientific Center of Roentgenoradiology ( Site 0559), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 0562), Moscow, Moscow
  - Omsk Clinical Oncology Dispensary ( Site 0568), Omsk, Omsk Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 0576), Samara, Samara Oblast
  - SBHI Leningrad Regional Oncology Dispensary ( Site 0588), Saint Petersburg, Sankt-Peterburg
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0570), Saint Petersburg, Sankt-Peterburg
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 0567), Saint Petersburg, Sankt-Peterburg
  - Tomsk National Scientific Medical Center of Russian Academy of Science ( Site 0579), Tomsk, Tomsk Oblast
- South Korea (5):
  - Chonnam National University Hwasun Hospital ( Site 0174), Hwasun Gun, Jeonranamdo
  - National Cancer Center ( Site 0176), Goyang-si, Kyonggi-do
  - Asan Medical Center ( Site 0171), Songpagu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 0173), Seoul
  - Samsung Medical Center ( Site 0172), Seoul
- Spain (9):
  - Instituto Catalan de Oncologia - ICO ( Site 0330), L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Tauli ( Site 0335), Sabadell, Barcelona
  - Hospital San Pedro de Alcantara ( Site 0326), Cáceres, Extremadura
  - Hospital Josep Trueta ( Site 0321), Girona, Gerona
  - Hospital Quiron Madrid ( Site 0325), Pozuelo de Alarcón, Madrid
  - Hospital del Mar ( Site 0333), Barcelona
  - Hospital General Universitari Vall d Hebron ( Site 0334), Barcelona
  - Hospital Clinic ( Site 0323), Barcelona
  - Hospital Universitario Virgen de la Victoria ( Site 0337), Málaga
- Taiwan (5):
  - National Cheng Kung University Hospital ( Site 0134), Tainen, Tainan
  - China Medical University Hospital ( Site 0132), Taichung
  - Taichung Veterans General Hospital ( Site 0133), Taichung
  - National Taiwan University Hospital ( Site 0131), Taipei
  - Taipei Veterans General Hospital ( Site 0135), Taipei
- United Kingdom (7):
  - University Hospitals Bristol NHS Foundation Trust ( Site 0530), Bristol, Bristol, City of
  - Cambridge University Hospitals NHS Trust ( Site 0540), Cambridge, Cambridgeshire
  - Torbay Hospital ( Site 0532), Torquay, Devon
  - Royal Marsden Hospital ( Site 0526), Sutton, England
  - Musgrove Park Hospital ( Site 0537), Taunton, England
  - University of North Midlands NHS Foundation Trust ( Site 0527), Stoke-on-Trent, Staffordshire
  - Mount Vernon Cancer Centre ( Site 0536), Northwood

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Antonarakis ES, Park SH, Goh JC, Shin SJ, Lee JL, Mehra N, McDermott R, Sala-Gonzalez N, Fong PC, Greil R, Retz M, Sade JP, Yanez P, Huang YH, Begbie SD, Gafanov RA, De Santis M, Rosenbaum E, Kolinsky MP, Rey F, Chiu KY, Roubaud G, Kramer G, Sumitomo M, Massari F, Suzuki H, Qiu P, Zhang J, Kim J, Poehlein CH, Yu EY. Pembrolizumab Plus Olaparib for Patients With Previously Treated and Biomarker-Unselected Metastatic Castration-Resistant Prostate Cancer: The Randomized, Open-Label, Phase III KEYLYNK-010 Trial. J Clin Oncol. 2023 Aug 1;41(22):3839-3850. doi: 10.1200/JCO.23.00233. Epub 2023 Jun 8. PMID 37290035
- [Derived] Mehra N, Antonarakis ES, Park SH, Goh JC, McDermott R, Sala Gonzalez N, Fong PC, Greil R, De Santis M, Yanez PE, Huang YH, Begbie SD, Rey F, Kramer G, Suzuki H, Saretsky TL, Ghate SR, Cui Y, Hosius C, Yu EY. Patient-reported Outcomes in KEYLYNK-010: Pembrolizumab Plus Olaparib Versus Abiraterone or Enzalutamide for Participants with Biomarker-unselected, Previously Treated Metastatic Castration-resistant Prostate Cancer. Eur Urol Oncol. 2025 Aug;8(4):1030-1040. doi: 10.1016/j.euo.2025.04.018. Epub 2025 Jul 19. PMID 40685311
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26344&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to the next-generation hormonal agent monotherapy (NHA) arm received one of two NHA treatments, per protocol.
Groups:
- Pembrolizumab + Olaparib: Participants received olaparib 600 mg as two 150 mg oral tablets twice daily (BID) continuously until progression PLUS on Day 1 of each 21-day cycle, pembrolizumab 200 mg by intravenous (IV) infusion for up to 35 cycles (approximately 2 years).
- Next-generation Hormonal Agent Monotherapy (NHA): Participants received a single NHA of either abiraterone acetate (participants previously treated with enzalutamide) 1000 mg as two 500 mg or four 250 mg oral tablets once daily (QD) PLUS prednisone or prednisolone 10 mg as one 5 mg tablet BID until progression OR participants received enzalutamide (participants previously treated with abiraterone acetate) 160 mg as four 40 mg oral tablets or capsules OR two 80 mg tablets QD until progression.
Period: Overall Study
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Started | 529 | 264
Treated | 526 | 256
Completed | 0 | 0
Not Completed | 529 | 264
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Death | 368 | 174
Not completed — Physician Decision | 5 | 1
Not completed — Sponsor decision | 149 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA) | Total
Number analyzed (Participants) | 529 | 264 | 793
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.9 (7.4) | 69.1 (7.3) | 69.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 529 | 264 | 793
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 32 | 103
  Not Hispanic or Latino | 441 | 219 | 660
  Unknown or Not Reported | 17 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 102 | 59 | 161
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 4 | 5
  White | 419 | 199 | 618
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 1 | 5
Measurable Response Evaluation Criteria in Solid Tumors Version 1.1 Disease Status at Baseline [Count of Participants; unit: Participants] — Measurable disease at baseline is defined as having disease that is Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)-measurable lesions per blinded independent central review (BICR).
  Participants
    RECIST Measurable: Yes | 244 | 119 | 363
    RECIST Measurable: No | 285 | 145 | 430
Prior Use of NHA Treatment [Count of Participants; unit: Participants] — Prior use of NHA treatment was defined as prior treatment with Abiraterone only, Enzalutamide only, or Abiraterone and Enzalutamide.
  Participants
    Abiraterone only | 289 | 143 | 432
    Enzalutamide only | 240 | 120 | 360
    Abiraterone and Enzalutamide | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death due to any cause. The nonparametric Kaplan-Meier method was used to estimate the survival curves.
Time Frame: Up to ~31 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | 15.8 [14.6 to 17.0] | 14.6 [12.6 to 17.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Treatment difference in survival assessed by the stratified log-rank test stratified by measurable disease status and prior NHA treatment; Test type: Superiority; p = 0.2616, Log Rank; One-sided p-value based on log-rank test stratified by measurable disease status and prior NHA treatment; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.77 to 1.14] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by measurable disease status and prior NHA treatment

2. Primary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: rPFS is defined as the time from randomization to the first documented progressive disease (PD) per PCWG-modified RECIST 1.1 based on BICR or death due to any cause, whichever occurred first. Per PCWG-modified RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions or ≥2 new bone lesions was also considered PD. PCWG-modified RECIST is similar to RECIST 1.1 with the exception that a confirmation assessment of PD (>4 weeks after the initial PD) is required for participants who remain on treatment following a documented PD per RECIST 1.1 and PCWG rules include new bone lesions. The rPFS per PCWG-modified RECIST as assessed by BICR for all participants is presented. The nonparametric Kaplan-Meier method was used to estimate the survival curves.
Time Frame: Up to ~26 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | 4.4 [4.2 to 6.0] | 4.2 [4.0 to 6.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Treatment difference in rPFS assessed by the stratified log-rank test stratified by measurable disease status and prior NHA treatment; Test type: Superiority; p = 0.5544, Log Rank; One-sided p-value based on log-rank test stratified by measurable disease status and prior NHA treatment; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.82 to 1.25] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Initiation of the First Subsequent Anticancer Therapy (TFST)
Description: TFST is the time from randomization to initiation of the first subsequent anticancer therapy defined as the first anti-cancer treatment not part of the study arm for a given participant, or death, whichever occurs first. The nonparametric Kaplan-Meier method was used to estimate the survival curves.
Time Frame: Up to ~26 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | 7.2 [6.7 to 8.1] | 5.7 [5.0 to 7.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in TFST; Hazard Ratio (HR) = 0.86, 95% CI [0.71 to 1.03] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions per RECIST 1.1 and no evidence of disease (NED) bone scan) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1 and Non-PD, non-evaluable (NE), or NED bone scan or CR with non-PD or NE bone scan.) The percentage of participants who experienced CR or PR as assessed by BICR is presented.
Time Frame: Up to ~31 months
Population: All randomized participants who had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 244 | 119
Percentage of Participants | 16.8 [12.3 to 22.1] | 5.9 [2.4 to 11.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in ORR; Difference in percentage = 10.9, 95% CI 2-sided [4.0 to 17.1]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per PCWG-modified RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of ≥ 2 new bone lesions is also considered PD. DOR as assessed by BICR is presented.
Time Frame: Up to ~26 months
Population: All randomized participants who experience a confirmed CR or PR and had measurable disease at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 41 | 7
Months | 8.1 [6.2 to 14.1] | 8.5 [5.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

6. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression is defined as the time from randomization to PSA progression. PSA progression date is defined as the date of:
  1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, OR 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline. The nonparametric Kaplan-Meier method was used to estimate the survival curves.
Time Frame: Up to ~31 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | 3.3 [3.0 to 3.5] | 3.5 [3.2 to 4.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in time to PSA progression; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.89 to 1.38] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to First Symptomatic Skeletal-Related Event (SSRE)
Description: SSRE is defined as the time from randomization to the first symptomatic skeletal-related event, defined as whichever occurs first:
  * First use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms;
  * Occurrence of new symptomatic pathologic bone fracture (vertebral or nonvertebral);
  * Occurrence of spinal cord compression; or
  * Tumor-related orthopedic surgical intervention
Time Frame: Up to ~31 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | NA [NA to NA] — NA = Lower limit, median, and upper limit were not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [NA to NA] — NA = Lower limit, median, and upper limit were not reached at time of data cut-off due to insufficient number of responding participants with relapse.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in SSRE; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.38 to 0.78] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to Radiographic Soft Tissue Progression
Description: Time to radiographic soft tissue progression is defined as the time from randomization to radiographic soft tissue progression per soft tissue rule of PCWG-modified RECIST 1.1. Progression is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Time to radiographic soft tissue progression as assessed by BICR is presented.
Time Frame: Up to ~31 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 529 | 264
Months | 10.3 [8.3 to 12.3] | 6.4 [6.1 to 10.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in time to radiographic soft tissue progression; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 1.00] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Time to Pain Progression (TTPP)
Description: TTPP is defined as the time from randomization to pain progression as determined by Item 3 of the Brief Pain Inventory Short Form (BPI-SF) and by the Analgesic Quantification Algorithm (AQA) score.
  Pain progression is defined as:
  1. For participants who are asymptomatic at baseline, a ≥2-point change from baseline in the average (4-7 days) BPI-SF item 3 score at 2 consecutive visits OR initiation of opioid use for pain
  2. For participants who are symptomatic at baseline (average BPI-SF Item 3 score >0 and/or currently taking opioids), a ≥2-point change from baseline in the average BPI-SF Item 3 score and an average worst pain score ≥4 and no decrease in average opioid use (≥1-point decrease in AQA score from a starting value of 2 or higher) OR any increase in opioid use at 2 consecutive follow-up visits.
  Participants who had more than 2 consecutive visits that were not evaluable for pain progression were censored at the last evaluable assessment.
Time Frame: Up to ~31 months
Population: All participants who have at least 1 assessment available and have received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 504 | 246
Months | 13.5 [9.7 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 12.0 [10.1 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of responding participants with relapse.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Next-generation Hormonal Agent Monotherapy (NHA); Test type: Other — Treatment difference in TTPE; p = 0.3643, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.72 to 1.26] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an adverse event are presented.
Time Frame: Up to ~55 months
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 526 | 256
Participants | 518 | 238

11. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE are presented.
Time Frame: Up to ~1461 Days
Population: All randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
Number analyzed (Participants) | 526 | 256
Participants | 90 | 11

ADVERSE EVENTS:
Time Frame: For All-Cause Mortality: from allocation up to ~55 months. For AEs from start of treatment up to ~55 months.
Description: All-cause mortality: All allocated participants. AEs: All allocated participants who received ≥1 dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs. The next-generation hormonal agent monotherapy interventions are considered standard of care (SOC).
Arm/Group | Pembrolizumab + Olaparib | Next-generation Hormonal Agent Monotherapy (NHA)
All-Cause Mortality (participants affected / at risk) | 372/529 | 178/264
Serious Adverse Events (participants affected / at risk) | 179/526 | 59/256
Other Adverse Events (participants affected / at risk) | 495/526 | 215/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Olaparib (N=526) | Next-generation Hormonal Agent Monotherapy (NHA) (N=256)
Anaemia (Blood and lymphatic system disorders) | 20 (22) | 3 (3)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 9 (9) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 4 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (2) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (15) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Prostatitis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Septic shock (Infections and infestations) | 5 (5) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (12) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 5 (5) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (4) | 4 (4)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (5) | 2 (3)
Urinary tract obstruction (Renal and urinary disorders) | 5 (5) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Olaparib (N=526) | Next-generation Hormonal Agent Monotherapy (NHA) (N=256)
Anaemia (Blood and lymphatic system disorders) | 272 (327) | 36 (38)
Hypothyroidism (Endocrine disorders) | 54 (55) | 4 (4)
Constipation (Gastrointestinal disorders) | 108 (124) | 44 (47)
Diarrhoea (Gastrointestinal disorders) | 103 (135) | 21 (25)
Nausea (Gastrointestinal disorders) | 223 (280) | 47 (51)
Vomiting (Gastrointestinal disorders) | 92 (149) | 18 (20)
Asthenia (General disorders) | 95 (109) | 27 (29)
Fatigue (General disorders) | 188 (200) | 66 (67)
Oedema peripheral (General disorders) | 48 (51) | 14 (16)
Pyrexia (General disorders) | 52 (61) | 7 (8)
Urinary tract infection (Infections and infestations) | 26 (33) | 13 (16)
Alanine aminotransferase increased (Investigations) | 29 (30) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 40 (49) | 10 (10)
Blood alkaline phosphatase increased (Investigations) | 35 (38) | 25 (28)
Blood creatinine increased (Investigations) | 47 (57) | 6 (6)
Weight decreased (Investigations) | 71 (74) | 15 (15)
Decreased appetite (Metabolism and nutrition disorders) | 155 (178) | 46 (53)
Arthralgia (Musculoskeletal and connective tissue disorders) | 99 (122) | 37 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 85 (95) | 45 (52)
Bone pain (Musculoskeletal and connective tissue disorders) | 35 (43) | 26 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (36) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 (40) | 23 (31)
Dizziness (Nervous system disorders) | 44 (53) | 9 (9)
Dysgeusia (Nervous system disorders) | 31 (32) | 3 (3)
Headache (Nervous system disorders) | 29 (36) | 13 (19)
Insomnia (Psychiatric disorders) | 24 (26) | 13 (14)
Haematuria (Renal and urinary disorders) | 27 (35) | 11 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (57) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (44) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 37 (47) | 3 (3)
Hot flush (Vascular disorders) | 11 (11) | 15 (15)
Hypertension (Vascular disorders) | 31 (37) | 31 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03834519/Prot_SAP_002.pdf